CLINICAL TRIAL: NCT03901053
Title: Comparative Effect of Commercially Available Custom Dynamic Orthoses (CDOs)
Brief Title: Ankle Foot Orthosis Comparative Effect
Acronym: AFOCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jason Wilken (Other)
Collaborators: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency); Walter Reed National Military Medical Center (U.S. Federal Agency); Henry M. Jackson Foundation for the Advancement of Military Medicine (Other); Center for Veterans Research and Education (Other); University of Delaware (Other); Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor-Investigator, Jason Wilken, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 201901829; CDMRP-OP170060 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2019-03-25; First posted 2019-04-03 (Actual); Results first posted 2025-10-31 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-10

CONDITIONS: Foot Injuries and Disorders
Keywords: Ankle Foot Orthoses; Carbon Fiber; Gait; Adult; Biomechanics; Materials Testing; Physical Performance
MeSH Terms: conditions — Foot Injuries; Disease

STUDY DESIGN:
Intervention Model Description: Participants will be cast, fit, and tested with each device in question (Reaktiv and PhatBrace AFO). Participants will be randomized to one of two arms (AB or BA) to maximize the likelihood of similarity between groups with respect to a range of anthropometric, demographic and injury related factors. We will use block randomization in groups of 4 to achieve equal randomization between groups over time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- AB (Experimental): Participants in this arm will receive the Reaktiv AFO made by FabTech Systems LLC first, then the PhatBrace AFO by Bio-Mechanical Composites Inc. second.
  Interventions: Device: Reaktiv AFO; Device: PhatBrace AFO
- BA (Experimental): Participants in this arm will receive the PhatBrace AFO by Bio-Mechanical Composites Inc. first, then the Reaktiv AFO made by FabTech Systems LLC second.
  Interventions: Device: Reaktiv AFO; Device: PhatBrace AFO

INTERVENTIONS:
Device: Reaktiv AFO — This device is a carbon fiber ankle foot orthosis (brace) that contacts the foot and lower leg. It consists of a foot plate that is designed to protect the foot, a carbon fiber strut on the back that stores and returns energy, and a cuff that goes below the knee. It has a custom geometry and alignment that is specific to the individual.
Device: PhatBrace AFO — Although lighter and thinner than the Reaktiv it has a similar overall design. The posterior strut is typically longer and the footplate is thinner, more compliant and less customized. Further, the device is formed into a single piece.

SUMMARY:
The proposed effort is designed to support evidence-based practice and optimal care by evaluating how the form, fit and function of two commercially available carbon fiber custom fit braces (Orthoses) influences outcomes following extremity injury. Early data suggests that custom fit carbon fiber braces can significantly improve function following severe lower leg injuries. The proposed study will provide evidence that can be used by clinicians to guide their practice, including care for service members, veterans and civilians who have experienced a high-energy traumatic injury to their lower leg.

DETAILED DESCRIPTION:
In this research study, adult participants who have sustained a below-the-knee traumatic injury greater than two years ago and are still experiencing deficits including weakness and/or immobility will be assigned to one of two brace sequences (AB or BA). Participants will be randomized to a particular sequence, with an equal chance of getting either order. Participants will be evaluated under 4 conditions: no device, standard of care, and 2 carbon fiber custom dynamic orthoses (CDO), the Reaktiv device from FabTech Systems and the PhatBrace by Bio-Mechanical Composites Inc. Participants will be tested with no device and standard of care at baseline, after 3 months of accommodation to the Reaktiv, and 3 months of accommodation to the PhatBrace. A series of study measures will be performed. The physical performance measures will incorporate tests of agility, balance, speed and lower limb power. Questionnaires will be used to evaluate participant's perceived comfort and smoothness, pain, preference, and semi-structured interviews will be used to fully capture the perspective of the participant. A motion capture system will be used to evaluate walking mechanics, allowing comparisons between conditions. Lower limb forces and body motion will be assessed using computerized motion capture and force plates in the floor, as individuals walk over-ground. Small reflective markers placed on the participant's skin and force measuring plates in the floor will be used. The investigators will also complete mechanical testing of the devices and collect demographic and descriptive data.

ELIGIBILITY:
Inclusion Criteria:

* Ages: 18-65
* Sustained a function limiting, below the knee, traumatic lower leg injury that occurred greater than two years ago
* Weakness of ankle plantarflexors (<4/5 on MMT), limited pain free ankle motion (DF<10deg or PF<20deg), mechanical pain with loading onto hindfoot/midfoot/forefoot (>4/10 on verbal numeric pain rating scale), ankle or hindfoot fusion or candidate for ankle or hindfoot fusion, AND/OR a candidate for amputation secondary to ankle/foot impairment
* Ability to walk 50 feet without using a cane or crutch
* Ability to walk at a slow to moderate pace
* Able to read and write in English and provide written informed consent

Exclusion Criteria:

* Pain > 8/10 while walking
* Ankle weakness as a result of spinal cord injury or central nervous system pathology
* Require a knee stabilizing device (i.e. Knee-Ankle Foot Orthosis or Knee Orthosis) to perform daily activities
* Surgery on study limb anticipated in the next 6 months
* Medical or psychological conditions that would preclude functional testing (ex. severe traumatic brain injury, heart condition, clotting disorder, lung condition, stroke, vestibular disorder)
* Nerve, muscle, bone, or other condition limiting function of the contralateral extremity
* BMI greater than 45
* Visual or hearing impairment that limit walking ability or limit the ability to comply with instructions given during testing
* Pregnancy- Per participant self-report. Due the expected small number of pregnant individuals and resulting inability to account for its effect on resulting outcomes participants will be withdrawn from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason M. Wilken, PT, PhD, Principal Investigator — University of Iowa
Locations (3):
- United States (3):
  - University of Iowa, Iowa City, Iowa
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Minneapolis VA Health Care System, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Four (4) of the participants in this study failed the post-informed consent screening checklist, and were excluded form the study before being assigned to either group. The fifty (50) eligible participants were randomized to one of the two groups.
Groups:
- Reaktiv, PhatBrace: Participants in this arm will receive the Reaktiv AFO made by FabTech Systems LLC first, then the PhatBrace AFO by Bio-Mechanical Composites Inc. second.
  Reaktiv AFO: This device is a carbon fiber ankle foot orthosis (brace) that contacts the foot and lower leg. It consists of a foot plate that is designed to protect the foot, a carbon fiber strut on the back that stores and returns energy, and a cuff that goes below the knee. It has a custom geometry and alignment that is specific to the individual.
  PhatBrace AFO: Although lighter and thinner than the Reaktiv it has a similar overall design. The posterior strut is typically longer and the footplate is thinner, more compliant and less customized. Further, the device is formed into a single piece.
- PhatBrace, Reaktiv: Participants in this arm will receive the PhatBrace AFO by Bio-Mechanical Composites Inc. first, then the Reaktiv AFO made by FabTech Systems LLC second.
  Reaktiv AFO: This device is a carbon fiber ankle foot orthosis (brace) that contacts the foot and lower leg. It consists of a foot plate that is designed to protect the foot, a carbon fiber strut on the back that stores and returns energy, and a cuff that goes below the knee. It has a custom geometry and alignment that is specific to the individual.
  PhatBrace AFO: Although lighter and thinner than the Reaktiv it has a similar overall design. The posterior strut is typically longer and the footplate is thinner, more compliant and less customized. Further, the device is formed into a single piece.
Period: Overall Study
Arm/Group | Reaktiv, PhatBrace | PhatBrace, Reaktiv
Started | 25 | 25
Completed | 12 | 14
Not Completed | 13 | 11
Not completed — Lost to Follow-up | 6 | 2
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Unsatisfactory Device | 1 | 2
Not completed — No longer meets study criteria | 1 | 3
Not completed — Subject's Medical Status | 0 | 1
Not completed — Screening Failure | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants completed study activities in each of the experimental conditions in a randomized order (Reaktiv, PhatBrace; PhatBrace Reaktiv)
Groups:
- Total: Total of all reporting groups
Arm/Group | Reaktiv, PhatBrace | PhatBrace, Reaktiv | Total
Number analyzed (Participants) | 12 | 14 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 13 | 25
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.3 (10.4) | 44.5 (10.8) | 41.7 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 8 | 10 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 10 | 13 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 13 | 23
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: PROMIS Patient Reported Outcomes for Physical Function
Description: The Patient Reported Outcome Information System (PROMIS) physical function Computer Adaptive Test (CAT) is a computerized assessment measuring physical function. It is scored using a T-score in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. In a given PROMIS domain, a T-score above 50 represents more of the measured variable than the population average.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Reaktiv: Reaktiv AFO: This device is a carbon fiber ankle foot orthosis (brace) that contacts the foot and lower leg. It consists of a foot plate that is designed to protect the foot, a carbon fiber strut on the back that stores and returns energy, and a cuff that goes below the knee. It has a custom geometry and alignment that is specific to the individual.
- PhatBrace: PhatBrace AFO: Although lighter and thinner than the Reaktiv it has a similar overall design. The posterior strut is typically longer and the footplate is thinner, more compliant and less customized. Further, the device is formed into a single piece.
Arm/Group | Reaktiv | PhatBrace
Number analyzed (Participants) | 26 | 26
score on a scale | 44.78 (6.01) | 45.02 (8.35)

2. Primary Outcome: PROMIS Patient Reported Outcomes for Pain Interference
Description: The Patient Reported Outcome Information System (PROMIS) pain interference Computer Adaptive Test (CAT) is a computerized assessment measuring pain interference. It is scored using a T-score in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. In a given PROMIS domain, a T-score above 50 represents more of the measured variable than the population average.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Reaktiv | PhatBrace
Number analyzed (Participants) | 26 | 26
T-score | 55.22 (6.30) | 53.49 (6.52)

3. Primary Outcome: Activities-Specific Balance Confidence (ABC)
Description: The Activities-Specific Balance Confidence (ABC) scale provides a standardized evaluation of balance confidence across a range of common daily tasks. Higher scores indicate more confidence, with 0 = no confidence and 100 = full confidence.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Reaktiv | PhatBrace
Number analyzed (Participants) | 26 | 26
units on a scale | 76.37 (19.66) | 76.92 (18.92)

4. Primary Outcome: Satisfaction With Device (OPUS - CSD)
Description: Satisfaction with device will be assessed using the Orthotics Prosthetics Users' Survey Satisfaction With Device Score (11-55). Higher scores indicate a better outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reaktiv | PhatBrace
Number analyzed (Participants) | 26 | 26
score on a scale | 35.88 (6.13) | 36.04 (8.06)

5. Primary Outcome: Modified Socket Comfort Score (Comfort)
Description: Comfort scores range from 0 = most uncomfortable to 10 = most comfortable.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reaktiv | PhatBrace
Number analyzed (Participants) | 26 | 26
score on a scale | 7.12 (2.10) | 7.12 (1.93)

6. Primary Outcome: Modified Socket Comfort Score (Comfort and Smoothness)
Description: Smoothness scores range from 0 = least smooth to 10 = most smooth.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reaktiv | PhatBrace
Number analyzed (Participants) | 26 | 26
score on a scale | 7.65 (1.92) | 7.46 (2.06)

7. Primary Outcome: Numerical Pain Rating Scale
Description: Pain will be assessed using a standard 11-point numerical pain rating scale, in which 0 = no pain and 10 = worst pain imaginable.
Time Frame: 3 months
Population: One participant failed to complete in-person physical performance measures in the PhatBrace condition, and their reported numerical pain rating was unable to be collected as a result.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reaktiv | PhatBrace
Number analyzed (Participants) | 26 | 25
score on a scale | 1.85 (2.03) | 1.68 (1.75)

8. Primary Outcome: Participant Device Preference
Description: The participant will rank order their preference for the Reaktiv and Phatbrace on a questionnaire.
Time Frame: After 3 months of accomodation with the final device (Crossover study)
Measure: Count of Participants; unit: Participants
Arm/Group | Reaktiv | PhatBrace
Number analyzed (Participants) | 26 | 26
Participants | 10 | 16

9. Primary Outcome: Four-square Step Test (4SST- Timed)
Description: The 4SST is a standardized timed test of balance and agility. Measured in seconds with lower scores indicating better balance and agility.
Time Frame: 3 months
Population: One participant did not complete in-person physical performance measures in the PhatBrace condition, and their four-square step test time was unable to be collected as a result.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Reaktiv | PhatBrace
Number analyzed (Participants) | 26 | 25
Seconds | 7.39 (1.72) | 7.06 (1.78)

10. Primary Outcome: Self-selected Walking Velocity (SSWV - Timed)
Description: SSWV will be assessed using the timed 10 meter walk test. Measured in seconds.
Time Frame: 3 months
Population: One participant did not complete in-person physical performance measures in the PhatBrace condition, and their self-selected walking velocity was unable to be collected as a result.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Reaktiv | PhatBrace
Number analyzed (Participants) | 26 | 25
Seconds | 4.46 (0.58) | 4.49 (0.60)

11. Primary Outcome: 10 Meter Shuttle Run (10M Shuttle - Timed)
Description: The 10 meter shuttle run is a well-established timed measure of speed. Measured in seconds.
Time Frame: 3 months
Population: One participant did not complete in-person physical performance measures in the PhatBrace condition, and their 10 meter shuttle run was unable to be collected as a result.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Reaktiv | PhatBrace
Number analyzed (Participants) | 26 | 25
Seconds | 19.05 (5.81) | 19.05 (6.41)

12. Primary Outcome: Ankle Joint Power
Description: Peak ankle joint moment (W/kg) during gait.
Time Frame: 3 months
Population: One participant did not complete the in-person biomechanics collection in the PhatBrace condition, and their ankle joint power was unable to be collected as a result.
Measure: Mean (Standard Deviation); unit: W/kg
Arm/Group | Reaktiv | PhatBrace
Number analyzed (Participants) | 26 | 25
W/kg | 1.43 (0.17) | 1.29 (0.27)

13. Primary Outcome: Center of Pressure Velocity Timing
Description: Timing of peak center of pressure velocity (percent stance) during gait.
Time Frame: 3 months
Population: One participant did not complete the in-person biomechanics collection in the PhatBrace condition, and their center of pressure velocity was unable to be collected as a result.
Measure: Mean (Standard Deviation); unit: percent of gait cycle
Arm/Group | Reaktiv | PhatBrace
Number analyzed (Participants) | 26 | 25
percent of gait cycle | 25.81 (12.69) | 15.11 (8.83)

14. Primary Outcome: Center of Pressure Velocity Magnitude
Description: Magnitude of peak center of pressure velocity (m/s) during gait.
Time Frame: 3 months
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Reaktiv | PhatBrace
Number analyzed (Participants) | 26 | 25
m/s | 0.89 (0.29) | 0.75 (0.21)

15. Secondary Outcome: PROMIS Patient Reported Outcomes for Satisfaction With Participation in Social Activities
Description: The Patient Reported Outcome Information System (PROMIS) satisfaction with participation in social activities Computer Adaptive Test (CAT) is a computerized assessment measuring satisfaction with participation in social activities. It is scored using a T-score in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. In a given PROMIS domain, a T-score above 50 represents more of the measured variable than the population average.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Reaktiv | PhatBrace
Number analyzed (Participants) | 26 | 26
T-score | 49.39 (7.58) | 48.42 (7.22)

16. Secondary Outcome: Paffenbarger Physical Activity Questionnaire
Description: Participants will report their physical activity using the Paffenbarger Physical Activity Questionnaire. Average hours of vigorous activity completed during the week and during the weekend will be recorded separately. Participants completed this questionnaire at the beginning of the study prior and reported baseline physical activity without wearing either CDO.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Reaktiv, PhatBrace | PhatBrace, Reaktiv
Number analyzed (Participants) | 12 | 14
Hours
  Average on weekday | 2.17 (2.25) | 1.66 (1.81)
  Average on weekend | 1.75 (2.09) | 2.39 (2.37)

17. Secondary Outcome: Ankle Joint Moment
Description: Peak ankle joint moment (Nm/kg) during gait.
Time Frame: 3 months
Population: One participant did not complete the in-person biomechanics collection in the PhatBrace condition, and their ankle joint moment was unable to be collected as a result.
Measure: Mean (Standard Deviation); unit: Nm/kg
Arm/Group | Reaktiv | PhatBrace
Number analyzed (Participants) | 26 | 25
Nm/kg | 1.43 (0.17) | 1.29 (0.27)

18. Other Pre Specified Outcome: PROMIS Patient Reported Outcomes for Pain Behavior
Description: The Patient Reported Outcome Information System (PROMIS) pain behavior Computer Adaptive Test (CAT) is a computerized assessment measuring pain behavior. It is scored using a T-score in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. In a given PROMIS domain, a T-score above 50 represents more of the measured variable than the population average.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Reaktiv | PhatBrace
Number analyzed (Participants) | 26 | 26
T-score | 55.22 (5.60) | 54.45 (7.79)

19. Other Pre Specified Outcome: PROMIS Patient Reported Outcomes for Depression
Description: The Patient Reported Outcome Information System (PROMIS) depression Computer Adaptive Test (CAT) is a computerized assessment measuring depression. It is scored using a T-score in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. In a given PROMIS domain, a T-score above 50 represents more of the measured variable than the population average.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Reaktiv | PhatBrace
Number analyzed (Participants) | 26 | 26
T-score | 48.24 (9.72) | 48.35 (8.86)

20. Other Pre Specified Outcome: PROMIS Patient Reported Outcomes for Satisfaction With Participation in Social Roles
Description: The Patient Reported Outcome Information System (PROMIS) satisfaction with participation in social roles Computer Adaptive Test (CAT) is a computerized assessment measuring satisfaction with participation in social roles. It is scored using a T-score in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. In a given PROMIS domain, a T-score above 50 represents more of the measured variable than the population average.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Reaktiv | PhatBrace
Number analyzed (Participants) | 26 | 26
T-score | 49.37 (8.56) | 48.70 (7.48)

21. Other Pre Specified Outcome: Satisfaction With Services (OPUS - CSS)
Description: Satisfaction with services will be assessed using the Orthotics Prosthetics Users' Survey Satisfaction With Services Score (10-50). Higher scores indicate a better outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reaktiv | PhatBrace
Number analyzed (Participants) | 26 | 26
score on a scale | 40.04 (8.47) | 38.65 (8.75)

22. Other Pre Specified Outcome: Sit to Stand 5 Times (STS5 - Timed)
Description: STS5 is a well-established timed measure of lower limb muscle strength and power. Participants are instructed to stand up and sit down 5 times as fast as possible.
Time Frame: 3 months
Population: One participant did not complete in-person physical performance measures in the PhatBrace condition, and their sit-to-stand time was unable to be collected as a result.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Reaktiv | PhatBrace
Number analyzed (Participants) | 26 | 25
Seconds | 8.94 (2.20) | 8.82 (2.55)

23. Other Pre Specified Outcome: Timed Stair Ascent (TSA - Timed)
Description: The timed stair ascent test is a measure of mobility, agility, and lower limb muscle strength. Participants are instructed to ascend a flight of 12 steps as quickly and safely as possible while contacting every step.
Time Frame: 3 months
Population: One participant did not complete in-person physical performance measures in the PhatBrace condition, and timed stair ascent was unable to be collected as a result.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Reaktiv | PhatBrace
Number analyzed (Participants) | 26 | 25
Seconds | 5.82 (2.97) | 5.43 (2.60)

ADVERSE EVENTS:
Time Frame: Study participants were asked to indicate any adverse events throughout the duration of each study visit. After completion of the study participants were also asked to call or email the research team if any adverse events related to the study occurred after the study visit (up to ~12 months after the visit).
Arm/Group | Reaktiv | PhatBrace
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-08): https://cdn.clinicaltrials.gov/large-docs/53/NCT03901053/Prot_SAP_000.pdf